CLINICAL TRIAL: NCT03341091
Title: The Effects of Simplified 10-step Tai-chi Programme on the Motor Performance and Fall Prevention of Community-dwelling Older People With Dementia: a Pilot Cluster Randomized Control Trial
Brief Title: Effects of Tai-chi Programme on Mobility of People With Dementia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4-ZZFT
Record Dates: First submitted 2017-11-08; First posted 2017-11-14 (Actual); Last update posted 2017-11-14 (Actual); Status verified 2017-11

CONDITIONS: Accidental Falls
Keywords: Tai-chi; Dementia; Dyad approach; Fall prevention; Mobility
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: A two-arm parallel (single-blinded) cluster randomised controlled trial involves two groups of participants (Tai-chi and the control group). Four community health centers that provide dementia care services were recruited through convenience sampling and each was viewed as one cluster and was randomised to either the Tai-chi or the control group, based on computer-generated random numbers. So during the trial, participants in one group receive Tai-chi group programme "in parallel" to participants in the other group, who took part in group recreational activities and continue their usual lifestyles and levels of physical activity.
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who was blinded to group allocation assessed the participants' motor performance variables.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tai-chi group (Experimental): 16-week 10-step simplified Tai-chi programme.
  Two 1-hour sessions of centre-based Tai-chi training and a minimum of three 30-minute Tai-chi sessions at home on a weekly basis.
  Interventions: Other: Tai-chi group
- Control group (No Intervention): Group recreational activities and continue their usual lifestyles and levels of physical activity as usual for 16 weeks.
  Two 1-hour sessions of group recreational activities on a weekly basis.

INTERVENTIONS:
Other: Tai-chi group — The Tai-chi group received a 16-week 10-step simplified Tai-chi training programme in which additional measures were implemented to enhance participants' engagement.
  Arms: Tai-chi group

SUMMARY:
This study evaluates the feasibility and the preliminary effects of a simplified 10-step Tai-chi programme (a dyadic approach) on the mobility performance of people with mild to moderate dementia.

Four community health centres were recruited and each was randomised to either the intervention group (Tai-chi) or the control group. Tai-chi group received a 16-week 10-step simplified Tai-chi training programme in which additional measures were implemented to enhance participants' engagement. The control group took part in group recreational activities organized by the community centres.

It was hypothesized that the Tai-chi group would outperform the control group regarding their mobility performance.

DETAILED DESCRIPTION:
Four community health centres that provide dementia care services were recruited through convenience sampling. Each was viewed as one cluster and was randomized to either the Tai-chi or the control group, based on computer-generated random numbers prepared by an independent statistician.

Participants allocated to the Tai-chi group took part in the 16-week 10-step simplified Tai-chi programme, which was derived from the traditional Yang style and has been proven to be effective in enhancing older people's balance and mobility. Each week, the dyads attended two 1-hour sessions of centre-based Tai-chi training and practised at least three 30-minute Tai-chi sessions at home. Additional measures targeted cognitively impaired people were implemented to promote engagement, including the adoption of multiple sensory cues, slow and relaxed practice, a dyadic approach, and positive emotional motivation techniques.

Participants allocated to the control group took part in group recreational activities such as watching movies or listening to music, which was organized by the community centres with similar frequency and duration of the Tai-chi sessions that were organized for the Tai-chi group. The control group participants were instructed to continue their usual lifestyles and levels of physical activity.

ELIGIBILITY:
Inclusion Criteria (for participants with dementia):

* community-dwelling older people aged > 60 years;
* able to walk independently with no walking aid or no more than a single point stick for at least 10 minutes to ensure their mobility was good enough for taking part in the Tai-chi training;
* formally diagnosed with a form of dementia;
* classified with mild to moderate severity of dementia, assessed by the Montreal Cognitive Assessment 5-minute scale with a cut-off score at the 16th percentile according to participants' age and education; and
* able to identify a caregiver who was willing to work as an exercise partner for their Tai-chi practice.

Inclusion Criteria (for caregivers):

* adults aged > 18;
* living with the participants or actively involved in their daily care;
* sufficiently mobile to be able to take part in the Tai-chi training together with the participants; and
* willing to work as an exercise partner with the participants and monitor and encourage them to practice Tai-chi at home.

Exclusion Criteria (for participants and caregivers):

if at the time of and three months before recruitment, they

* had any diseases that might severely affect their balance and coordination, such as Parkinson's disease or myasthenia gravis;
* were hospitalized due to acute illnesses such as myocardial infarction, stroke or hip fracture, or had major surgeries;
* reported that they regularly performed moderately intensive exercise, such as hiking or Tai-chi, for more than 2 hours per week;
* had terminal illnesses such as cancer and were in palliative care; or
* had severe visual or hearing impairment.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-11-01 (Actual); Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Enrollment date
  The number of dyads who provided consent to join the study over the eligible dyads
Attrition rate | At the end of the 16-week programme
  The attrition rate was indicated by the percentage of dyads withdrawing from the study
Participants' adherence to practising Tai-chi at home and in the training sessions | Throughout the 16-week programme
  Exercise adherence (Tai-chi group only) was assessed by both the exercise diaries and training session attendance. Caregivers were instructed to record participants' adherence in terms of the frequency and duration of their Tai-chi home practice in a weekly exercise diary.
Occurrence of adverse events such as falls | Throughout the 16-week programme and during the training sessions
  Any adverse events at home were recorded.

SECONDARY OUTCOMES:
Time measured in the Timed-up-and-Go test | Baseline, 8th week and 16th week from baseline
  The Timed-up-and-Go test assess mobility of the participants. The time taken by participants to execute the tasks - stand up from a standard chair, walk three meters, turn around, walk back to the chair and sit down - was recorded in seconds.
Time measured in the Timed Chair Stand test | Baseline, 8th week and 16th week from baseline
  Timed Chair Stand test assesses functional lower limb muscle strength of the participant. Each participant was instructed to stand up fully and sit down five times as quickly as possible. The time needed to complete this task was recorded.
Length measured by the Functional Reach test | Baseline, 8th week and 16th week from baseline
  Functional Reach test assessed the dynamic bilateral stance balance of the participants. Participants stood beside a wall with their dominant arm raised to 90 degrees. They were then instructed to lean forward as far as possible, with the hand remaining at shoulder level. The Functional Reach score was the additional reach of the raised hand from the starting position in centimeters
Number of steps recorded in the Step Test | Baseline, 8th week and 16th week from baseline
  The Step Test assesses the dynamic single leg standing balance of the participants. Participants stood with their feet parallel and apart. They were instructed to place one whole foot onto the 5 centimetre-high block in front of them and then return it fully back down to the floor repeatedly as fast as possible, for 15 seconds. Each leg was tested separately, and performance on the side with the least number of steps was the recorded result.
Focus interview groups | 17th week from baseline
  Feedback from participants and their caregivers was collected by focus group within two weeks of completing the Tai-chi programme
Menorah Park Engagement Scale | every week of the 16-week Tai-chi programme
  The engagement of participants with dementia when attending the Tai-chi training sessions was assessed by four items extracted from the Menorah Park Engagement Scale. The four items are constructive engagement, passive engagement, self/other engagement, and non-engagement. Each item was rated on a three-point Likert scale (i.e., 0 = "not observed", 1 = "up to half the observation", and 2 = "more than half of the observation"). In addition, Engagement was also rated by the Tai-chi master on a 4-item scale (i.e. engagement during class, following proper steps, satisfaction with participants' learning progress, and satisfaction with participants' performance) based on the Tai-chi instructor's in-class observation. Each item was quantified on a 10-point Likert scale, with higher scores representing a greater degree of engagement.

CONTACTS AND LOCATIONS:
Overall Officials: Yat-wa Justina Liu, Principal Investigator — The Hong Kong Polytechnic University
Locations (2):
- Hong Kong (2):
  - Caritas Hong Kong - Services for the Elderly, Hong Kong
  - H.K.S.K.H. Lok Man Alice Kwok Integrated Service Centre, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the names of all participants including the caregivers will be replaced by reference codes. The data collected will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 3 years after the completion of this research.

REFERENCES:
- [Background] Kim SH. Risk factors for severe injury following indoor and outdoor falls in geriatric patients. Arch Gerontol Geriatr. 2016 Jan-Feb;62:75-82. doi: 10.1016/j.archger.2015.10.003. Epub 2015 Oct 22. PMID 26553485
- [Background] Global Burden of Disease Study 2013 Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 301 acute and chronic diseases and injuries in 188 countries, 1990-2013: a systematic analysis for the Global Burden of Disease Study 2013. Lancet. 2015 Aug 22;386(9995):743-800. doi: 10.1016/S0140-6736(15)60692-4. Epub 2015 Jun 7. PMID 26063472
- [Background] Taylor ME, Delbaere K, Close JC, et al. Managing falls in older patients with cognitive impairment. Aging Health 2012; 8: 573-588.
- [Background] Muir SW, Gopaul K, Montero Odasso MM. The role of cognitive impairment in fall risk among older adults: a systematic review and meta-analysis. Age Ageing. 2012 May;41(3):299-308. doi: 10.1093/ageing/afs012. Epub 2012 Feb 27. PMID 22374645
- [Background] Gillespie LD, Robertson MC, Gillespie WJ, Lamb SE, Gates S, Cumming RG, Rowe BH. Interventions for preventing falls in older people living in the community. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD007146. doi: 10.1002/14651858.CD007146.pub2. PMID 19370674
- [Background] Harling A and Simpson JP. A systematic review to determine the effectiveness of Tai Chi in reducing falls and fear of falling in older adults. Physical Therapy Reviews 2008; 13: 237-248.
- [Background] Logghe IH, Verhagen AP, Rademaker AC, Bierma-Zeinstra SM, van Rossum E, Faber MJ, Koes BW. The effects of Tai Chi on fall prevention, fear of falling and balance in older people: a meta-analysis. Prev Med. 2010 Sep-Oct;51(3-4):222-7. doi: 10.1016/j.ypmed.2010.06.003. Epub 2010 Jun 15. PMID 20558197
- [Background] Huang Y, Liu X. Improvement of balance control ability and flexibility in the elderly Tai Chi Chuan (TCC) practitioners: a systematic review and meta-analysis. Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):233-8. doi: 10.1016/j.archger.2014.10.016. Epub 2014 Nov 18. PMID 25497683
- [Background] Song R, Ahn S, So H, Lee EH, Chung Y, Park M. Effects of t'ai chi on balance: a population-based meta-analysis. J Altern Complement Med. 2015 Mar;21(3):141-51. doi: 10.1089/acm.2014.0056. Epub 2015 Feb 4. PMID 25650522
- [Background] Yao L, Giordani BJ, Algase DL, You M, Alexander NB. Fall risk-relevant functional mobility outcomes in dementia following dyadic tai chi exercise. West J Nurs Res. 2013 Mar;35(3):281-96. doi: 10.1177/0193945912443319. Epub 2012 Apr 19. PMID 22517441
- [Background] Liu-Ambrose T, Ahamed Y, Graf P, Feldman F, Robinovitch SN. Older fallers with poor working memory overestimate their postural limits. Arch Phys Med Rehabil. 2008 Jul;89(7):1335-40. doi: 10.1016/j.apmr.2007.11.052. PMID 18586136
- [Background] Shaw FE, Bond J, Richardson DA, Dawson P, Steen IN, McKeith IG, Kenny RA. Multifactorial intervention after a fall in older people with cognitive impairment and dementia presenting to the accident and emergency department: randomised controlled trial. BMJ. 2003 Jan 11;326(7380):73. doi: 10.1136/bmj.326.7380.73. PMID 12521968
- [Background] Close J, Ellis M, Hooper R, Glucksman E, Jackson S, Swift C. Prevention of falls in the elderly trial (PROFET): a randomised controlled trial. Lancet. 1999 Jan 9;353(9147):93-7. doi: 10.1016/S0140-6736(98)06119-4. PMID 10023893
- [Background] Meyer C, Hill S, Dow B, Synnot A, Hill K. Translating Falls Prevention Knowledge to Community-Dwelling Older PLWD: A Mixed-Method Systematic Review. Gerontologist. 2015 Aug;55(4):560-74. doi: 10.1093/geront/gnt127. Epub 2013 Nov 11. PMID 24218145
- [Background] Small JA. A new frontier in spaced retrieval memory training for persons with Alzheimer's disease. Neuropsychol Rehabil. 2012;22(3):329-61. doi: 10.1080/09602011.2011.640468. Epub 2012 Jan 24. PMID 22272562
- [Background] Burgener SC, Yang Y, Gilbert R, Marsh-Yant S. The effects of a multimodal intervention on outcomes of persons with early-stage dementia. Am J Alzheimers Dis Other Demen. 2008 Aug-Sep;23(4):382-94. doi: 10.1177/1533317508317527. Epub 2008 May 4. PMID 18453642
- [Background] Tsai PF, Chang JY, Beck C, Kuo YF, Keefe FJ. A pilot cluster-randomized trial of a 20-week Tai Chi program in elders with cognitive impairment and osteoarthritic knee: effects on pain and other health outcomes. J Pain Symptom Manage. 2013 Apr;45(4):660-9. doi: 10.1016/j.jpainsymman.2012.04.009. Epub 2012 Sep 24. PMID 23017610
- [Background] Lam LC, Chau RC, Wong BM, Fung AW, Lui VW, Tam CC, Leung GT, Kwok TC, Chiu HF, Ng S, Chan WM. Interim follow-up of a randomized controlled trial comparing Chinese style mind body (Tai Chi) and stretching exercises on cognitive function in subjects at risk of progressive cognitive decline. Int J Geriatr Psychiatry. 2011 Jul;26(7):733-40. doi: 10.1002/gps.2602. Epub 2010 Dec 9. PMID 21495078
- [Background] Yao L, Giordani B, Alexander NB. Developing a positive emotion-motivated Tai Chi (PEM-TC) exercise program for older adults with dementia. Res Theory Nurs Pract. 2008;22(4):241-55. PMID 19093662
- [Background] Chang JY, Tsai PF, Woods S, Beck C, Roberson PK, Rosengren K. Teaching Tai Chi to elders with osteoarthritis pain and mild cognitive impairment. Am J Recreat Ther. 2011 Winter;10(1):11-16. PMID 25242898
- [Background] Liu YW, Tsui CM. A randomized trial comparing Tai Chi with and without cognitive-behavioral intervention (CBI) to reduce fear of falling in community-dwelling elderly people. Arch Gerontol Geriatr. 2014 Sep-Oct;59(2):317-25. doi: 10.1016/j.archger.2014.05.008. Epub 2014 May 29. PMID 24953768
- [Background] Tinetti ME, Powell L. Fear of falling and low self-efficacy: a case of dependence in elderly persons. J Gerontol. 1993 Sep;48 Spec No:35-8. doi: 10.1093/geronj/48.special_issue.35. No abstract available. PMID 8409238
- [Background] Judge KS, Camp CJ and Orsulic-Jeras S. Use of Montessori-based activities for clients with dementia in adult day care: Effects on engagement. American Journal of Alzheimer's Disease 2000; 15: 42-46.
- [Background] Podsiadlo D, Richardson S. The timed "Up & Go": a test of basic functional mobility for frail elderly persons. J Am Geriatr Soc. 1991 Feb;39(2):142-8. doi: 10.1111/j.1532-5415.1991.tb01616.x. PMID 1991946
- [Background] Hatch J, Gill-Body KM, Portney LG. Determinants of balance confidence in community-dwelling elderly people. Phys Ther. 2003 Dec;83(12):1072-9. PMID 14640866
- [Background] Whitney SL, Wrisley DM, Marchetti GF, Gee MA, Redfern MS, Furman JM. Clinical measurement of sit-to-stand performance in people with balance disorders: validity of data for the Five-Times-Sit-to-Stand Test. Phys Ther. 2005 Oct;85(10):1034-45. PMID 16180952
- [Background] Duncan PW, Weiner DK, Chandler J, Studenski S. Functional reach: a new clinical measure of balance. J Gerontol. 1990 Nov;45(6):M192-7. doi: 10.1093/geronj/45.6.m192. PMID 2229941
- [Background] Hill KD, Bernhardt J, McGann AM, et al. A new test of dynamic standing balance for stroke patients: reliability, validity and comparison with healthy elderly. Physiotherapy Canada 1996; 48: 257-262.
- [Background] Hill K, Denisenko S, Miller K, et al. Clinical outcome measurement in adult neurological physiotherapy. Victoria: Australian Physiotherapy Association National Neurology Group 2005.
- [Background] Suttanon P, Hill KD, Dodd KJ, Said CM. Retest reliability of balance and mobility measurements in people with mild to moderate Alzheimer's disease. Int Psychogeriatr. 2011 Sep;23(7):1152-9. doi: 10.1017/S1041610211000639. Epub 2011 Apr 14. PMID 21489342
- [Background] Suttanon P, Hill KD, Said CM, Williams SB, Byrne KN, LoGiudice D, Lautenschlager NT, Dodd KJ. Feasibility, safety and preliminary evidence of the effectiveness of a home-based exercise programme for older people with Alzheimer's disease: a pilot randomized controlled trial. Clin Rehabil. 2013 May;27(5):427-38. doi: 10.1177/0269215512460877. Epub 2012 Nov 1. PMID 23117349
- [Derived] Liu JYW, Kwan RYC, Lai CK, Hill KD. A simplified 10-step Tai-chi programme to enable people with dementia to improve their motor performance: a feasibility study. Clin Rehabil. 2018 Dec;32(12):1609-1623. doi: 10.1177/0269215518786530. Epub 2018 Jul 4. PMID 29969916

DOCUMENTS (3):
  • Informed Consent Form (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03341091/ICF_000.pdf
  • Statistical Analysis Plan (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03341091/SAP_001.pdf
  • Study Protocol (2016-05-16): https://cdn.clinicaltrials.gov/large-docs/91/NCT03341091/Prot_002.pdf